CLINICAL TRIAL: NCT05963659
Title: The Effect of Nitrate on Cognitive Function in Alcohol Dependence Patients and the Potential Microbiota Mechanism.
Brief Title: Nitrate Modulates Cognitive Impairment Via Oral Microbiota.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Sixth Hospital (Other)
Responsible Party: Principal Investigator, Hongqiang Sun, Clinical Professor,Director, Peking University Sixth Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20230630
Record Dates: First submitted 2023-06-30; First posted 2023-07-27 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Microtia; Alcohol Dependence
Keywords: nitrate; oral microbiota; alcohol dependence
MeSH Terms: conditions — Congenital Microtia; Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group N (Experimental)
  Interventions: Dietary Supplement: nitrate-rich beetroot juice
- Group P (Placebo Comparator)
  Interventions: Dietary Supplement: nitrate-depleted beetroot juice

INTERVENTIONS:
Dietary Supplement: nitrate-rich beetroot juice — nitrate-rich beetroot juice, ~750 mg NO3- /d
  Arms: Group N
Dietary Supplement: nitrate-depleted beetroot juice — nitrate-depleted beetroot juice, ~1 mg NO3- /d
  Arms: Group P

SUMMARY:
Alcohol use is increasingly prevalent in modern society and is known to cause cognitive impairment and dysregulation of inflammatory responses. In the present study, the investigators want to perform a randomised controlled trials to test whether nitrate could change the oral microbiota and benefit the cognitive impairment in alcohol dependence patients. The investigators survey the oral bacterial communities in saliva samples of 70 alcohol dependent patients following 14 days of dietary inorganic nitrate (nitrate-rich beetroot juice, ~750 mg NO3- /d) and placebo (nitrate-depleted beetroot juice, ~1 mg NO3- /d) supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. Han nationality
2. Montreal Cognitive Assessment(MoCA) score >11
3. Diagnosis of alcohol dependence

Exclusion Criteria:

1. Past or current infectious disease
2. Past or current heart, brain, liver, kidney, and other severe diseases
3. Past or current metabolic diseases that can lead to abnormalities of the immune system, such as obesity (Body Mass Index > 30 kg/m2), diabetes, or rheumatoid arthritis
4. Past or current neurodegenerative diseases, such as Parkinson's disease
5. Use of steroidal and non-steroidal anti-inflammatory drugs, antibiotics, antioxidants, and immunosuppressive agents within two months of enrollment
6. Use of probiotics and probiotics every day for the first two months before enrollment
7. Previous or current DSM-IV diagnosis of schizophrenia, depression, anxiety disorder, bipolar disorder, mental retardation, dementia (excluding mild cognitive impairment, MCI), or substance dependence other than alcohol and nicotine
8. Irregular eating habits that affect the oral flora (except alcohol) in the previous two months
9. Current oral disease

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
Changes of Delayed Match to Sample Percent Correct (all delays) from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by DMS-PCAD (Delayed Match to Sample Percent Correct , all delays)
Changes of Spatial Working Memory Between Errors from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by SWM-BE (The Spatial Working Memory Between Errors )

SECONDARY OUTCOMES:
Changes of oral microbiota from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Saliva samples were used to test the composition of microbiota by 16S RNA sequencing.
Changes of gut microbiota from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Feces samples were used to test the composition of microbiota by 16S RNA sequencing.
Changes of Delayed Match to Sample Percent Correct (0 seconds delay) from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by Delayed Match to Sample Percent Correct (0 seconds delay)
Changes of Delayed Match to Sample Percent Correct (4 seconds delay) from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by Delayed Match to Sample Percent Correct (4 seconds delay)
Changes of Delayed Match to Sample Percent Correct (12 seconds delay) from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by Delayed Match to Sample Percent Correct (12 seconds delay)
Changes of Spatial Working Memory errors 4 boxes from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by The Spatial Working Memory errors 4 boxes
Changes of Spatial Working Memory errors 6 boxes from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by The Spatial Working Memory errors 6 boxes
Changes of Spatial Working Memory errors 8 boxes from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by The Spatial Working Memory errors 8 boxes
Changes of Intra-Extra Dimensional Set Shift test Stages Completed from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by The Intra-Extra Dimensional Set Shift test Stages Completed
Changes of Intra-Extra Dimensional Completed Stage Errors from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by The Intra-Extra Dimensional Completed Stage Errors
Changes of Cambridge Gambling Task Risk Adjustment Merged: Risk adjustment from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by Cambridge Gambling Task Risk Adjustment Merged: Risk adjustment
Changes of Cambridge Gambling Decision Making Quality Total Merged from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by Cambridge Gambling Decision Making Quality Total Merged
Changes of Cambridge Gambling Delay Aversion Total from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by Cambridge Gambling Delay Aversion Total
Changes of Reaction Time Median Five-Choice Movement Time from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by Reaction Time Median Five-Choice Movement Time
Changes of Reaction Time Median Five-Choice Reaction Time from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by Reaction Time Median Five-Choice Reaction Time
Changes of Rapid Visual Information Processing test Probability of False Alarm from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by the Rapid Visual Information Processing test Probability of False Alarm
Changes of Rapid Visual Information Processing test A prime from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by the Rapid Visual Information Processing test A prime
Changes of Rapid Visual Information Processing test Median Response Latency from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  Test by the Rapid Visual Information Processing test Median Response Latency
Changes of nitrate levels in serum from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  The collected serum samples were used to test the levels of nitrate and nitrite by High Performance Liquid Chromatography \ HPLC
Changes of nitrite levels in serum from baseline to post-intervention | baseline and post-intervention(two weeks after baseline test)
  The collected serum samples were used to test the levels of nitrate and nitrite by High Performance Liquid Chromatography \ HPLC

OTHER OUTCOMES:
Systolic and diastolic blood pressure | baseline and post-intervention (two weeks after baseline test)
  Test by blood pressure monitor
Cytokine Tumor Necrosis Factor-a in serum | baseline and post-intervention(two weeks after baseline test)
  The collected serum samples were used to test the levels of TNF-a by Enzyme-Linked Immunosorbent Assay
The blood biochemical related parameters includes liver enzymes (alanine aminotransferase and aspartate aminotransferase) | baseline and post-intervention (two weeks after baseline test)
  The collected venous blood were sent to the department of clinical laboratory and the investigators recorded the laboratory report.
The blood biochemical related parameters blood fat (cholesterol, triglycerides, low density lipoprotein and high density lipoprotein | baseline and post-intervention (two weeks after baseline test)
  The collected venous blood were sent to the department of clinical laboratory and the investigators recorded the laboratory report.
Cytokine Interleukin-1b in serum | baseline and post-intervention(two weeks after baseline test)
  The collected serum samples were used to test the levels of IL-1b by Enzyme-Linked Immunosorbent Assay
Cytokine Interleukin-6 in serum | baseline and post-intervention (two weeks after baseline test)
  The collected serum samples were used to test the levels of IL-6 by Enzyme-Linked Immunosorbent Assay
Cytokine Interleukin-10 in serum | baseline and post-intervention (two weeks after baseline test)
  The collected serum samples were used to test the levels of IL-10 by Enzyme-Linked Immunosorbent Assay

CONTACTS AND LOCATIONS:
Overall Officials: Hongqiang Sun, Principal Investigator — Peking University Sixth Hospital; Liangjun Pang, Study Chair — Anhui mental health central
Locations (1):
- Anhui mental health center, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No